CLINICAL TRIAL: NCT00250731
Title: Improving Diabetes Outcomes: a Couples Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Syracuse University (Other)
Responsible Party: Paula M. Trief, PhD/Professor, SUNY Upstate Medical University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DK06799501A2
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes
Keywords: diabetes; relationship; social support; behavior change; telemedicine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Telephone support and behavior change for couples
  Interventions: Behavioral: telephone support and behavior change
- 2 (Active Comparator): Telephone support and behavior change for individuals
  Interventions: Behavioral: telephone support and behavior change
- 3 (Placebo Comparator): Limited diabetes self-management education
  Interventions: Other: Diabetes self-management education

INTERVENTIONS:
Behavioral: telephone support and behavior change — Diabetes self-management education provided over the telephone either for individuals or couples
  Arms: 1; 2
Other: Diabetes self-management education — Limited diabetes self-management education provided over the telephone, serves as an enhanced usual care control intervention
  Arms: 3

SUMMARY:
Research has shown that diabetes affects both the patient and family, and that support from family and partners helps diabetes patients manage their illness better. However, diabetes programs rarely involve the partner. This is a study to develop and test an intervention that helps partners and patients who have type 2 diabetes better support each other. The intervention will be delivered over the telephone to reach more people. Our hypothesis is that an intervention that targets the couple has a greater effect on health and well-being of patients than one that targets the individual patient alone.

DETAILED DESCRIPTION:
Research has shown that diabetes affects both the patient and family, and that support from family and partners helps diabetes patients manage their illness better. However, diabetes programs rarely involve the partner. This is a pilot proposal to develop and test an intervention that aims to both enlist the support of partners of diabetes patients, and enhance and improve the quality of that support. We believe that the intervention will help the relationship and also will have a positive impact on medical (e.g.,blood sugar control), behavioral (e.g., increased exercise, better diet) and emotional (e.g., depression) outcomes. The intervention will be implemented by telephone, in order to enhance the project's ability to reach a broader sample of patients.Forty-five couples will be recruited in which one partner has type 2 diabetes. After initial testing and basic diabetes education, they will be assigned to one of three comparison groups. For those in the intervention groups they will participate in 11 telephone contacts with a diabetes educator and a counselor and will receive education about diabetes, behavior change, emotional issues/couples communication, and problem solving techniques. A manual will include readings, structured homework assignments, and self-monitoring logs. They will be re-tested 2 weeks and 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* greater than 21 years of age.
* diagnosed with type 2 diabetes for at least 1 year.
* have no severe complications (on dialysis, blindness, amputations, history of stroke)
* able to speak, read and hear English.
* married or cohabiting for > 1 year.
* have a telephone.

Exclusion Criteria:

* have a diagnosed psychiatric disorder.
* refuse audiotaping or other study procedures.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
blood glucose control (hemoglobin A1c) | 2 and 14 weeks post
blood pressure | 2 and 14 weeks post
diabetes regimen adherence | at 2 and 14 weeks post

SECONDARY OUTCOMES:
lipids | at 2 and 14 weeks post intervention
weight/BMI | at 2 and 14 weeks post intervention
food habits | at 2 and 14 weeks post intervention
activity habits | at 2 and 14 weeks post intervention
health-related quality of life | at 2 and 14 weeks post
relationship quality | at 2 and 14 weeks post intervention
diabetes self-efficacy | at 2 and 14 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Trief, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- State University of New York Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Garfield SA, Malozowski S, Chin MH, Narayan KM, Glasgow RE, Green LW, Hiss RG, Krumholz HM; Diabetes Mellitus Interagency Coordinating Committee (DIMCC) Translation Conference Working Group. Considerations for diabetes translational research in real-world settings. Diabetes Care. 2003 Sep;26(9):2670-4. doi: 10.2337/diacare.26.9.2670. No abstract available. PMID 12941736
- [Background] Delamater AM, Jacobson AM, Anderson B, Cox D, Fisher L, Lustman P, Rubin R, Wysocki T; Psychosocial Therapies Working Group. Psychosocial therapies in diabetes: report of the Psychosocial Therapies Working Group. Diabetes Care. 2001 Jul;24(7):1286-92. doi: 10.2337/diacare.24.7.1286. PMID 11423517
- [Background] Fisher L, Chesla CA, Bartz RJ, Gilliss C, Skaff MA, Sabogal F, Kanter RA, Lutz CP. The family and type 2 diabetes: a framework for intervention. Diabetes Educ. 1998 Sep-Oct;24(5):599-607. doi: 10.1177/014572179802400504. PMID 9830956
- [Background] Kiecolt-Glaser JK, Newton TL. Marriage and health: his and hers. Psychol Bull. 2001 Jul;127(4):472-503. doi: 10.1037/0033-2909.127.4.472. PMID 11439708
- [Background] Trief PM, Himes CL, Orendorff R, Weinstock RS. The marital relationship and psychosocial adaptation and glycemic control of individuals with diabetes. Diabetes Care. 2001 Aug;24(8):1384-9. doi: 10.2337/diacare.24.8.1384. PMID 11473074
- [Background] Trief PM, Wade MJ, Britton KD, Weinstock RS. A prospective analysis of marital relationship factors and quality of life in diabetes. Diabetes Care. 2002 Jul;25(7):1154-8. doi: 10.2337/diacare.25.7.1154. PMID 12087013
- [Background] Trief PM, Ploutz-Snyder R, Britton KD, Weinstock RS. The relationship between marital quality and adherence to the diabetes care regimen. Ann Behav Med. 2004 Jun;27(3):148-54. doi: 10.1207/s15324796abm2703_2. PMID 15184090
- [Derived] Trief P, Sandberg JG, Ploutz-Snyder R, Brittain R, Cibula D, Scales K, Weinstock RS. Promoting couples collaboration in type 2 diabetes: the diabetes support project pilot data. Fam Syst Health. 2011 Sep;29(3):253-61. doi: 10.1037/a0024564. PMID 21744962